CLINICAL TRIAL: NCT01170286
Title: Epicutaneous Immunotherapy (EPIT) for Peanut Allergy: A Randomized, Double-Blind, Placebo-Controlled Phase 1 Safety Study in Adult and Pediatric Subjects
Brief Title: Safety of Epicutaneous Immunotherapy for the Treatment of Peanut Allergy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: DBV Technologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PEP01.09
Record Dates: First submitted 2010-07-24; First posted 2010-07-27 (Estimated); Last update posted 2012-03-23 (Estimated); Status verified 2012-03

CONDITIONS: Peanut Allergy
Keywords: Food allergy; Immediate hypersensitivity; Whole peanut extract; Allergenic product; Specific Immunotherapy; Epicutaneous Immunotherapy (EPIT); Safety
MeSH Terms: conditions — Peanut Hypersensitivity; Food Hypersensitivity; Hypersensitivity, Immediate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DBV712 Viaskin (Experimental): The experimental arm is composed of subjects treated with whole peanut extract on an epicutaneous delivery system (Viaskin patch)
  Interventions: Biological: Whole peanut extract
- Placebo Viaskin (Placebo Comparator): The placebo arm is composed of subjects treated with a placebo formulation on an epicutaneous delivery system (Viaskin patch)
  Interventions: Biological: Placebo formulation

INTERVENTIONS:
Biological: Whole peanut extract — Four different doses of whole peanut extract expressed as micrograms (mcg) of peanut proteins (20, 100, 250, 500 mcg) and two different dosing regimen (epicutaneous application for 24 hours every 24 hours and epicutaneous application for 48 hours every 48 hours) will be tested for determination of the maximum tolerated dose during a 2-week treatment period.
  Other Names: DBV712 Viaskin
  Arms: DBV712 Viaskin
Biological: Placebo formulation — Matching placebo at two different dosing regimen (epicutaneous application for 24 hours every 24 hours and epicutaneous application for 48 hours every 48 hours) will be tested in parallel to the peanut proteins doses for determination of the maximum tolerated dose during a 2-week treatment period.
  Other Names: Placebo Viaskin
  Arms: Placebo Viaskin

SUMMARY:
The purpose of this phase 1b study is to evaluate the safety and tolerability of repeated epicutaneous applications of peanut proteins using a patch delivery system (Viaskin device) in peanut allergic subjects.

DETAILED DESCRIPTION:
Peanut allergy is a common allergy in the United States, with a prevalence in the general population as high as 1%. So far, there is no approved treatment of peanut allergy. Peanut allergy management is based on strict peanut avoidance and injectable epinephrine after the allergic systemic reactions have started. Specific Immunotherapy methods currently available have shown some limitations in their use because of safety issues. Hence, there is an important unmet medical need for efficient and safe treatment of peanut allergy.

DBV Technologies has developed an epicutaneous delivery system, called Viaskin, a method based on delivering precise quantity of the allergen on the upper layers of the skin. Avoiding contact between the allergen and the bloodstream should confer to epicutaneous immunotherapy (EPIT) a higher level of safety as systemic reactions should be circumvented.

The aim of this phase 1b study is to evaluate the safety and tolerability of the epicutaneous immunotherapy method in subjects allergic to peanut. The trial will randomize 110 participants. Four doses of peanut proteins, 20 mcg, 100 mcg, 250 mcg and 500 mcg will be repeatedly delivered on the skin by dose escalation in consecutive cohorts of 5 subjects, starting with the lowest dose. In each cohort of 5, 4 subjects will receive peanut proteins and one will receive placebo in a blinded manner. For each dose, the peanut proteins will be applied on the skin either every day or every other day. The total duration of the treatment for each subject is 2 weeks. Firstly, adult subjects (18 to 50 years) with a history of non-severe anaphylaxis to peanut (Grade ≤3) will enroll and safety information be reviewed. If there are no major concerns, adolescent cohorts (12 to 17 years) with history of non-severe anaphylaxis to peanut will then enroll and safety again be reviewed. If there are no concerns, then child cohorts (6 to 11 years) with history of non-severe anaphylaxis to peanut will finally enroll.

Also, after the safety review of the treated adult non-severe cohorts is satisfactorily performed, adult subjects with a history of severe anaphylaxis to peanut (Grades 4 or 5) will enroll and dose escalation will undergo.

For the safety review, all the following parameters will be checked at each patient visit: physical examination, vital signs, skin examination, lab values, PEF values. FEV1, skin prick test to peanut and peanut-specific IgE values will also be determined at screening and end of treatment visits.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female age 6 to 50 years at enrollment, any race, and any ethnicity.
* Physician-diagnosed peanut allergy or convincing history of peanut allergy regardless of the degree of the reaction. Subjects with history of severe anaphylaxis to peanuts (Grades 4 or 5 with dyspnea, cyanosis, hypoxia, hypotension, or neurological compromise) can be enrolled only after assessment of the safety of DBV712 Viaskin in subjects with historic non-severe anaphylaxis (Grade≤3).
* A peanut-specific IgE measured by ImmunoCAP >0.7 kU/L for all subjects and a positive skin prick test to peanut with a wheal diameter >8 mm for all non-severe subjects. A skin prick test to peanut for severe subjects will be performed only if deemed necessary by the investigator.
* Use of an effective method of contraception by females of childbearing potential and agreement to continue to practice an acceptable method of contraception for the duration of their participation in the study. Women who have had a hysterectomy or tubal ligation at least 6 months prior to the screening visit or who have been post-menopausal for at least 1 year prior to the screening visit are not considered to be of childbearing potential.
* Ability to perform spirometry maneuvers in accordance with the American Thoracic Society guidelines (1994).
* Able to understand the protocol and willing to comply with all study requirements during participation in the study.
* Provide signed informed consent and assent as appropriate.

Exclusion Criteria:

* Participation in a study using an investigational new drug in the last 30 days prior to the screening visit.
* Participation in any interventional study for the treatment of food allergy in the past 6 months prior to the screening visit.
* Pregnancy or lactation.
* Allergy or known hypersensitivity to the Viaskin patch or adhesives.
* Severe or poorly controlled atopic dermatitis or generalized eczema.
* FEV1 value <80% predicted or any clinical features of moderate or severe persistent asthma at baseline and treated by doses greater than high daily doses of inhaled corticosteroids (as defined in dosing tables from the 2007 NHLBI guidelines).
* Use of steroid medications in the following manners: history of daily oral steroid dosing for >1 month during the past year, or burst oral steroid course in the past 6 months, or >1 burst oral steroid course in the past year, prior to the screening visit. Use of oral steroids as described above after the screening visit and before randomization will render the subject non eligible for randomization.
* Asthma requiring 1 or more hospitalization(s) in the past year or >1 emergency department visit in the past 6 months, prior to the screening visit. Occurrence of asthma in these conditions after the screening visit and before randomization will render the subject non eligible for randomization.
* Use of omalizumab or immunomodulatory or biologic therapy in the past year prior to the screening visit.
* Use of nontraditional forms of allergen immunotherapy (such as oral immunotherapy or sublingual immunotherapy) in the past year prior to the screening visit.
* Use of subcutaneous immunotherapy other than a stable maintenance dose for less than a year prior to the screening visit.
* Use of beta-blockers, angiotensin-converting enzyme inhibitors, or angiotensin-receptor blockers.
* Inability to discontinue antihistamines for at least 1 week to allow skin testing at the screening visit.
* History of alcohol or drug abuse.
* Uncontrolled hypertension.
* History of cardiovascular disease, arrhythmias, chronic lung disease, active eosinophilic gastrointestinal disease, malignancy, psychiatric illness, or any other medical or surgical conditions which, in the opinion of the investigator, place the subject at increased risk for participation in this study.
* Inability or unwillingness to sign informed consent or to provide assent (as appropriate).
* Inability to speak English, including caretakers of participants when the participant is a child.

Ages: 6 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2010-07; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Safety evaluation | Safety evaluation to be performed at each visit during the 2-week treatment and at the follow-up visit one week after the end of treatment.
  The primary outcome measure is safety and the subjects will undergo the following procedures: physical examination including patch application site examination for evaluation of any skin reaction, vital signs, blood and urine collection for blood and urine analysis, ECG, Peak Expiratory Flow and spirometry (FEV1).
  Adverse events, treatment-emergent adverse events, and serious adverse events will be classified according to severity, treatment relatedness, the system/organ class affected, and the countermeasures taken.

SECONDARY OUTCOMES:
Systemic reactions evaluation and treatment; treatment adherence | Safety evaluation to be performed at each visit during the 2-week treatment and at the follow-up visit one week after the end of treatment.
  Secondary outcomes:
  1. The proportion of subjects that experience systemic reactions such as urticaria, asthma and acute dyspnea, change in blood pressure, and digestive symptoms (vomiting, diarrhea) associated with experimental treatment versus placebo.
  2. The proportion of subjects requiring treatment for systemic reactions related to experimental treatment or placebo.
  3. Overall adherence to the study treatment

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - National Jewish Health, Denver, Colorado
  - CRI Worldwide, Willingboro, New Jersey
  - Duke University Medical Center, Durham, North Carolina
  - Aspen Clinical Research, Orem, Utah

REFERENCES:
- [Derived] Jones SM, Agbotounou WK, Fleischer DM, Burks AW, Pesek RD, Harris MW, Martin L, Thebault C, Ruban C, Benhamou PH. Safety of epicutaneous immunotherapy for the treatment of peanut allergy: A phase 1 study using the Viaskin patch. J Allergy Clin Immunol. 2016 Apr;137(4):1258-1261.e10. doi: 10.1016/j.jaci.2016.01.008. Epub 2016 Feb 24. No abstract available. PMID 26920463